CLINICAL TRIAL: NCT06305520
Title: Medical Device Pivotal Study to Evaluate the Efficacy and Safety of Injection With SkinPlus-HYAL Implant Lidocaine as Compared to RESTYLANE Lidocaine in Temporary Correction of Nasolabial Folds
Brief Title: Medical Device Pivotal Study to Injection With SkinPlus-HYAL Implant Lidocaine vs RESTYLANE Lidocaine in of Nasolabial Folds
Acronym: BPLUS-02
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bioplus (Industry)
Collaborators: Seoul National University Hospital (Other); Asan Medical Center (Other); Soonchunhyang University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPLUS-NASAL-02; CRIS NO. : KCT0008113 (Registry Identifier: The Clinical Research Information Service (CRIS) in KOREA)
Record Dates: First submitted 2024-03-01; First posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Nasal Disease; Nasal Surgery
Keywords: Nasolabial fold; Filler; Medical Device
MeSH Terms: conditions — Nose Diseases

STUDY DESIGN:
Intervention Model Description: Medical Device
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Medical Device (Experimental): Application of the investigational medical device (SkinPlus-HYAL Implant Lidocaine)
  Interventions: Device: Investigational medical device (SkinPlus-HYAL Implant Lidocaine)
- Active Comparator Medical Device (Active Comparator): Application of the control device (RESTYLANE Lidocaine)
  Interventions: Device: Active Comparator: Active Comparator Medical Device (RESTYLANE Lidocaine)

INTERVENTIONS:
Device: Investigational medical device (SkinPlus-HYAL Implant Lidocaine) — * In this investigation, the same subject receives both test and control treatments, one on each side of the nasolabial folds (matched pairs design).
  Arms: Investigational Medical Device
Device: Active Comparator: Active Comparator Medical Device (RESTYLANE Lidocaine) — * In this investigation, the same subject receives both test and control treatments, one on each side of the nasolabial folds (matched pairs design).
  Arms: Active Comparator Medical Device

SUMMARY:
Purpose : This investigation intends to demonstrate that the investigational device, SkinPlus-HYAL Implant Lidocaine, is non-inferior to the comparator device, RESTYLANE Lidocaine, in terms of temporary wrinkle reduction effect, safety, and injection site pain when applied on nasolabial folds in adults.

Design : 24-week efficacy and safety evaluation and additional 48-week long-term safety and efficacy evaluation with a multi-center, randomized, subject- & evaluator-blind, matched pairs, active controlled, none-inferiority, confirmatory design

Treatment Group: Application of the investigational medical device (SkinPlus-HYAL Implant Lidocaine) Control Group: Application of the comparator device (RESTYLANE Lidocaine)

Population: Number of subject 100

* In this investigation, the same subject receives both test and control treatments, one on each side of the nasolabial folds (matched pairs design).

ELIGIBILITY:
Inclusion Criteria:

* Men and women 19 years of age or older
* Seeking temporary improvement of bilateral nasolabial folds, with a Wrinkle Severity Rating Scale (WSRS) score of 3 or 4 (does not have to be the same on both sides)
* Agrees to discontinue all dermatologic procedures or treatments (fillers, botulinum toxin, laser treatments, chemical peels, surgery for cosmetic purposes, etc.) other than investigational device application, including facial wrinkle improvement
* Able to understand and follow instructions and able to participate in all periods of the investigation
* Made a voluntary decision to participate in this investigation and gave written informed consent

Exclusion Criteria:

* Took antithrombotic agents (except low-dose aspirin (100 mg, maximum 300 mg/day)) from 2 weeks before to 2 weeks after application of the investigational device; took vitamin E formulations or NSAID formulations from 1 week before to 1 week after application
* History of bleeding disorder in the past or at the time of screening
* CaHA (Calcium Hydroxyapatite) or PLLA (Poly L-Lactide) filler treatment at the site of application of the investigational medical device within 1 year before the screening date
* Has used or intends to use topical agents (steroids, retinoids: medicines only, excluding cosmetics) on the facial area within 4 weeks before the screening date or during the clinical trial period (however steroid ointments for therapeutic purposes may be used for a short period of time within 14 consecutive days).
* Used immunosuppressants, chemotherapeutic agents, or systemic corticosteroids within 12 weeks before the screening date.
* Received any anti-wrinkle or acne scar treatment within 24 weeks before the screening date.
* Received dermabrasion, skin resurfacing, or cosmetic surgery (including botulinum toxin injections) to the facial area within 24 weeks before the screening date
* Permanent skin augmentation implants such as hardened gel (Softform) or silicone in the facial area
* Skin diseases or wound infections in the facial area that would affect this investigation
* History of autoimmune disease
* Hypersensitivity to sodium hyaluronate
* History of streptococcal disease
* History of anaphylaxis or severe multiple allergies
* History of hypertrophic scars, hyperpigmentation or keloids
* Hypersensitivity to lidocaine or other amide local anesthetics
* Coagulation disorders
* Clinically significant disorders of the cardiovascular, digestive, respiratory, endocrine, or central nervous systems or a psychiatric illness that significantly affects this investigation
* Participated in another clinical investigation within 30 days before the screening date and received/applied an investigational drug/investigational medical device
* Female subjects of childbearing potential who do not agree to use a medically acceptable method of contraception* until 48 weeks after application of the investigational medical device in this investigation. (*Medically accepted methods of contraception include: condoms, oral contraception continued for at least 3 months, use of injectable or insertable contraceptives, intrauterine contraceptive devices, etc.)
* Pregnant or lactating women
* Used steroid medication for therapeutic purposes (immune diseases, musculoskeletal diseases, etc.) within 4 weeks prior to enrollment in the investigation, or plans to use steroid medication during the investigation period
* Used or intends to use functional cosmetics for wrinkle improvement within 4 weeks before participation in the investigation or during the investigation period
* In addition to the above, those who have clinical significant findings that are considered inappropriate for this investigation by the principal investigator or personnel in charge, based on medical judgment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Difference in the mean values of the Wrinkle Severity Rating Scale (WSRS) between the treatment and control groups as evaluated by an independent evaluator at 24 weeks after the application of the investigational medical device | 24 weeks
  Descriptive statistics (number of observed subjects, mean, standard deviation, median, minimum, and maximum) for WSRS scores assessed by independent evaluators at 24 weeks after clinical trial device application by treatment group are presented. If the upper limit of the 97.5% one-sided confidence interval by t-distribution is less than 0.29 for the difference between treatment groups (test-control), it is judged that the non-inferiority of the test group has been demonstrated compared to the control group.
  WSRS is a measure of wrinkles from a minimum of 0 to a maximum of 5, and the higher the score, the deeper the wrinkles.

SECONDARY OUTCOMES:
Difference in the mean values of the WSRS between the treatment and control groups as evaluated by the investigator at 8, 16, 24, and 48 weeks after device application | 8, 16, 24, 48 weeks
  Descriptive statistics of WSRS scores (number of observed subjects, mean, standard deviation, median, minimum, and maximum) evaluated by test subjects at 8, 16, 24, and 48 weeks after medical device application for each treatment group are presented and analyzed by Wilcoxon's rank sum test if there is a difference between the administration groups.
  WSRS is a measure of wrinkles from a minimum of 0 to a maximum of 5, and the higher the score, the deeper the wrinkles.
Difference in the mean Global Aesthetic Improvement Scale (GAIS) values between the treatment and control groups as evaluated by the investigator at weeks 8, 16, 24, and 48 of the first post-device application phase compared to before application | 8, 16, 24, 48 weeks
  Descriptive statistics of GAIS scores (number of observed subjects, mean, standard deviation, median, minimum, and maximum values) evaluated by test subjects at 8, 16, 24, and 48 weeks after medical device application are presented for each treatment group and analyzed by Wilcoxon's rank sum test if there is a difference between the administration groups.
  GAIS is satisfaction with device usage from a minimum of 0 to a maximum of 5 points, and the higher the score, the higher the satisfaction.
Difference in the mean values of the WSRS between the treatment and control groups as evaluated by an independent evaluator at 48 weeks after device application. | 48 weeks
  Descriptive statistics of WSRS scores (number of observed subjects, mean, standard deviation, median, minimum, and maximum) evaluated by test subjects at 8, 16, 24, and 48 weeks after medical device application for each treatment group are presented and analyzed by Wilcoxon's rank sum test if there is a difference between the administration groups.
  WSRS is a measure of wrinkles from a minimum of 0 to a maximum of 5, and the higher the score, the deeper the wrinkles.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongnogu, South Korea

IPD SHARING:
Plan to Share IPD: No